CLINICAL TRIAL: NCT00488865
Title: RexMedical- Option* Vena Cava Filter IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rex Medical (Industry)
Responsible Party: Lindsay Carter, Rex Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REX-US-2006-001
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2010-08-05 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Pulmonary Embolism
Keywords: increased risk for PE require caval interruption
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravascular Filter Device (Other)
  Interventions: Device: Intravascular Filter Device

INTERVENTIONS:
Device: Intravascular Filter Device — Vena cava filter which is implanted into the inferior vena cava of patients to prevent recurrent pulmonary embolism. The filter can be utilized as a permanent or retrievable device.

SUMMARY:
This study is designed to evaluate the safety and efficacy of the RexMedical Option* Vena Cava Filter in the treatment of patients who are at increased risk for Pulmonary Embolism and require caval interruption.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is at least 18 years of age
* Patient requires temporary or permanent caval interruption

Key Exclusion Criteria:

* Patient has pre-existing filter implanted in her/her vasculature or has undergone filter retrieval within 60 days prior to study device implant
* Patient is currently enrolled in another investigational device or drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Peninsula Surgical Specialists Medical Group, Inc., Burlingame, California
  - Christiana Care Health System, Newark, Delaware
  - George Washington University, Washington D.C., District of Columbia
  - Miami Cardiac & Vascular Institute, Miami, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - New York Presbyterian Hospital/Columbia, New York, New York
  - OHSU, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Johnson MS, Nemcek AA Jr, Benenati JF, Baumann DS, Dolmatch BL, Kaufman JA, Garcia MJ, Stecker MS, Venbrux AC, Haskal ZJ, Avelar RL. The safety and effectiveness of the retrievable option inferior vena cava filter: a United States prospective multicenter clinical study. J Vasc Interv Radiol. 2010 Aug;21(8):1173-84. doi: 10.1016/j.jvir.2010.04.004. Epub 2010 Jul 3. PMID 20598570

RESULTS

PARTICIPANT FLOW:
Groups:
- Option IVC Filter Device Placement: All participants in the study will have an Option IVC filter placed for the prevention of recurrent pulmonary embolism.
Period: Overall Study
Arm/Group | Option IVC Filter Device Placement
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Option IVC Filter Device Placement
Number analyzed (Participants) | 100
Age, Customized [Number; unit: participants]
  <18 years | 0
  >=18 years | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Success
Description: Placement Technical Success without subsequent pulmonary embolism, significant filter migration, symptomatic caval thrombosis or other complication requiring filter removal or invasive intervention to address condition.
Time Frame: up to 180 days
Population: The number of participants was determined per intention to treat (ITT).
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Option IVC Filter Device Placement
Number analyzed (Participants) | 100
Percent of Participants | 88 [81 to 100]

2. Secondary Outcome: Placement Technical Success
Description: Successful deployment of the filter at the intended placement level such that the filter is judged suitable by the Investigator for mechanical protection against pulmonary embolism.
Time Frame: Immediately post placement procedure
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Option IVC Filter Device Placement
Number analyzed (Participants) | 100
Percent of Participants | 100 [100 to 100]

3. Primary Outcome: Percentage of Participants With Retrieval Clinical Success
Description: Intact filter retrieval via percutaneous techniques from the vasculature without associated injury or damage to the vena cava requiring intervention.
Time Frame: upto 175 days
Population: The population for Option filter retrieval was based on intention to treat (ITT). Retrieval procedures were attempted in 39 of the 100 enrolled patients.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Option IVC Filter Device Placement
Number analyzed (Participants) | 39
Percent of Participants | 92 [81 to 100]

ADVERSE EVENTS:
Arm/Group | Option IVC Filter Device Placement
Serious Adverse Events (participants affected / at risk) | 65/100
Other Adverse Events (participants affected / at risk) | 73/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Option IVC Filter Device Placement (N=100)
Device/Procedure Related SAE (General disorders) | 13 (17)
Non Device/Procedure Related SAE (General disorders) | 62 (216)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Option IVC Filter Device Placement (N=100)
Device/Procedure Related AE (General disorders) | 16 (20)
Non Device/Procedure Related AE (General disorders) | 73 (338)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No